CLINICAL TRIAL: NCT05665543
Title: Increasing HPV Vaccination Coverage Among Pediatric, Adolescent, and Young Adult (PAYA) Cancer Survivors: A Multilevel Intervention
Brief Title: Increasing HPV Vaccination in Pediatric, Adolescent, and Young Adult (PAYA) Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021LS099
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cancer; HPV Associated Cancer
Keywords: HPV vaccine
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLAm App (Experimental): Participants will have access to Game based Learning Avatar navigated mobile (GLAm ) app and will receive the receive the quality improvement (QI) intervention plus the GLAm app.
  Interventions: Behavioral: GLAm app
- Usual care (No Intervention): Participants in the control group will not receive the access to the GLAm app. They will receive the quality improvement (QI) intervention only.

INTERVENTIONS:
Behavioral: GLAm app — Game-based Learning Avatar-navigated mobile (app) provides information on HPV infection susceptibility, risk of HPV-associated cancers, screening methods, and ways to overcome screening barriers. Users navigate the app using an avatar, and earn points for game components completed. The app prompts screening using text message reminders based on patient-entered information, and links to schedule cervical cancer screening. Completing cervical cancer screening earns an electronic badge visible to other users via an anonymous screen name and avatar.
  Arms: GLAm App

SUMMARY:
The primary objectives of this study are to increase HPV vaccination initiation and 3-dose completion among pediatric, adolescent, and young adult (PAYA) cancer survivors

DETAILED DESCRIPTION:
PAYA cancer survivors are 2.8 times more likely to develop a secondary human papillomavirus (HPV)-associated cancer than the general population. Unfortunately, HPV vaccination coverage among PAYA cancer survivors is even lower than that in the general population. Provision of adequate vaccine information and instructions for timing of vaccination post-treatment is associated with an increased intention to vaccinate. Nonetheless, research show a minority of cancer care teams specifically discuss HPV vaccination with PAYA cancer survivors and their caregivers. The purpose of this study is to test the efficacy of an oncologist- and clinic-level intervention and the additional effect of a patient-level app-based intervention to improve initiation and 3-dose completion of the HPV vaccine series.

ELIGIBILITY:
Inclusion Criteria:

* Current patient in the University of Minnesota CCSP clinic or the Children's Minnesota Long-Term Follow-up (LTFU) Program clinic.
* Patients seen in the CCSP clinic who do not have a history of cancer but who have received immunosuppressive therapy or HSCT for treatment of a hematologic disorder.
* Survivor of childhood cancer (defined as diagnosed with cancer at age 25 years or younger) who is currently 18-26 years of age OR a caregiver of a survivor of childhood cancer who is currently 9-17 years of age.
* 6+ months post-treatment; current treatment for graft-versus-host disease allowed
* No previous HPV vaccination or incomplete HPV vaccination (defined as <3 doses post-cancer therapy). Individuals who are unsure of their HPV vaccination status who are unable to find vaccination records per the procedures detailed in Section 5.2, EHR support will be eligible, in concordance with real-world clinical practice regarding HPV vaccination.

Exclusion Criteria:

* Previous completion of the HPV vaccination series. Those who are eligible for re-vaccination per the CDC guidelines will be encouraged by their oncologist to re-vaccinate, but will not be included in the QI study or RCT.
* Unable to read/write in English per self-report (only applies to participants in the RCT [Aim 2]).
* Pregnant at the time of enrollment or plans to become pregnant in the next year. Pregnancy test at the time of enrollment is not required if pregnancy not clinically suspected in concordance with clinical guidelines for HPV vaccine administration.
* Currently receiving treatment for cancer or hematologic disorder or plan for treatment within 12 months of enrollment; treatment for graft-versus-host disease allowed.
* Other contraindications to the HPV vaccine (e.g. history of immediate hypersensitivity reaction to any vaccine component, including yeast).

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 162 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Study enrollment | within 6 months of index clinic visit
  Number of participants who complete the 3-dose HPV vaccine series within 12 months of study enrollment.

SECONDARY OUTCOMES:
Change in HPV and HPV vaccination knowledge pre- and post-intervention | baseline and 1 year post survivorship clinic visit
  The change in knowledge is assessed through self reported surveys administered to participants
Number of participants intent to vaccinate against HPV | At the time of index clinic visit, baseline
  The number of participants with intent to vaccinate is assessed through self reported surveys administered to participants
Proportion of participants intending to vaccinate initiating and completing the vaccine series | 1 year post index clinic visit
  The Proportion of participants intending to vaccinate initiating and completing the vaccine series is measured through surveys and health record review
Demographics differences associated with vaccination status | 1 year post index clinic visit
  measure through health record review
Cancer occurrences associated with vaccination status | 1 year post index clinic visit
  measure through health record review
Treatment differences associated with vaccination status | 1 year post index clinic visit
  measure through health record review
Number of participants experiencing barriers to vaccination | 1 year post index clinic visit
  Survey measurement
Number of participants using and accepting the game based learning app | 1 year post index clinic visit
  Survey measurement
Concordance between reported and documented vaccination against HPV | 1 year post index clinic visit
  measured through surveys and health record review

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Teoh, MD, MS, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, the link between subjects' identifiable identification codes and their identifiable information will be destroyed per the AHC protocol at the time of data disposal. The original data records will be archived for 7 years (in accordance with data practices).